CLINICAL TRIAL: NCT01890109
Title: Randomized, Stratified, Parallel-group, Double-blind, Placebo-controlled, Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of AMG 334 in Women With Hot Flashes Associated With Menopause
Brief Title: Study of Erenumab (AMG 334) in Women With Hot Flashes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20120180
Record Dates: First submitted 2013-05-13; First posted 2013-07-01 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Vasomotor Symptoms; Hot Flashes
Keywords: Vasomotor symptoms; Hot Flashes; Menopause
MeSH Terms: conditions — Hot Flashes | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received a single dose of placebo administered by subcutaneous injection.
  Interventions: Drug: Placebo
- Erenumab (Experimental): Participants received a single dose of 70 mg erenumab administered by subcutaneous injection.
  Interventions: Biological: Erenumab

INTERVENTIONS:
Biological: Erenumab — Administered via subcutaneous injection.
  Other Names: AMG 334; Aimovig™
  Arms: Erenumab
Drug: Placebo — Administered via subcutaneous injection
  Arms: Placebo

SUMMARY:
The primary objective of this study was to evaluate the frequency of moderate to severe daily hot flashes 4 weeks after a single dose of erenumab (AMG 334) in women with hot flashes associated with menopause.

DETAILED DESCRIPTION:
This study will test the hypothesis that the vasodilation associated with capsaicin-induced dermal blood flow (DBF) provides a good model for the vasodilation associated with hot flashes; therefore erenumab doses that cause DBF inhibition will be safe and well tolerated, and will be effective in the reduction of the frequency and/or severity of HFs.

ELIGIBILITY:
Inclusion Criteria:

* female subjects with hot flashes associated with menopause between 45 and 65 years of age, inclusive, with no history or evidence of clinically relevant medical disorders as determined by the investigator in consultation with the Amgen physician.

Exclusion Criteria:

* History or evidence of clinically significant disorder (including psychiatric), condition or disease that, in the opinion of the Investigator or Amgen physician would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2014-03-11 (Actual); Study Completion 2014-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (7):
  - Research Site, San Diego, California
  - Research Site, Miami, Florida
  - Research Site, Winston-Salem, North Carolina
  - Eugene Andruczyk, Philadelphia, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Seattle, Washington

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 6 centers in the United States from 13 May 2013 to 11 March 2014.
  Screening included completion of a 7-day diary to record hot flashes.
Pre-assignment Details: Participants meeting the eligibility criteria were randomized in a 1:1 ratio to erenumab or placebo. Participants were stratified based on the average number of hot flashes per 24 hours during the screening period (≤ 11.5 or > 11.5).
Period: Overall Study
Arm/Group | Placebo | Erenumab
Started | 52 | 51
Received Study Treatment | 52 | 50
Completed | 51 | 46
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: Participants who received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Erenumab | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (4.8) | 55.6 (3.8) | 55.6 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 102
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 46 | 42 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Black or African American | 15 | 10 | 25
  Mixed Race | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  White | 36 | 36 | 72
Number of Hot Flashes at Baseline [Count of Participants; unit: Participants] — Baseline number of hot flashes is the average number of moderate or severe hot flashes per 24 hours from day -7 to day 1 predose.
  Participants
    ≤ 11.5 hot flashes/24 hours | 26 | 25 | 51
    > 11.5 hot flashes/24 hours | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Week 4 to Baseline Average Number of Daily Moderate to Severe Hot Flashes
Description: The severity of hot flashes was assessed by participants based on the following categories:
  * Mild: sensation of heat without sweating, mild flushing;
  * Moderate: sensation of heat, face flushed, slightly clammy, some sweating, able to continue activity, may want to remove layers of clothing or covers at night;
  * Severe: sensation of heat with more severe sweating, have to stop current activity, may have to change clothing.
  Baseline (BL) number of hot flashes is the average number of moderate or severe hot flashes per 24 hours from day -7 to day 1 predose based on geometric mean, and the week 4 number of hot flashes is the average number of moderate or severe hot flashes per 24 hours from day 21 to day 27 based on geometric mean.
  The ratio of week 4 to BL was used to assess change from BL to week 4 via a log transformation (log[week4/BL] = log[week4] - log[BL]), which was estimated using a repeated measures analysis. The ratio was obtained via an exponential back-transformation.
Time Frame: Baseline (days -7 to day 1 predose) and week 4 (days 21 to 27)
Population: All participants for whom at least 1 postdose hot flash response measure was recorded.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 52 | 50
ratio | 0.35 [0.24 to 0.50] | 0.38 [0.26 to 0.55]
Statistical Analysis 1: Comparison: Placebo vs Erenumab; Repeated measures analysis of covariance was performed on the log transformed ratio to baseline of the number of daily moderate to severe hot flashes. Independent variables included treatment, week, and the treatment-by-week interaction; subject served as a random effect; and the log transformed baseline number of daily moderate to severe hot flashes was used as a covariate; Test type: Superiority; p = 0.723, Repeated Measures Analysis of Covariance; Least Square Geometric Mean Ratio = 1.10, 95% CI 2-sided [0.66 to 1.83]

2. Secondary Outcome: Ratio of Week 4 to Baseline Daily Hot Flash Severity Score
Description: The daily severity score was calculated according to the following:
  (Number of mild hot flashes * 1) + (number of moderate hot flashes * 2) + (number of severe hot flashes * 3).
  The baseline daily hot flash severity score is the geometric mean daily hot flash severity score from day -7 to day 1 predose, and the week 4 daily hot flash severity score is the geometric mean daily hot flash severity score from day 21 to day 27.
  The ratio of week 4 to baseline (week 4 / baseline) was used to assess change from baseline to week 4 via a log transformation (log[week4/BL] = log[week4] - log[baseline]), which was estimated using a repeated measures analysis. The ratio was obtained via an exponential back-transformation.
Time Frame: Baseline (days -7 to day 1 predose) and week 4 (days 21 to 27)
Population: All participants for whom at least 1 postdose hot flash response measure was recorded.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 52 | 50
ratio | 0.40 [0.29 to 0.53] | 0.45 [0.33 to 0.61]
Statistical Analysis 1: Comparison: Placebo vs Erenumab; Repeated measures analysis of covariance was performed on the log transformed ratio to baseline of the daily hot flash severity score. Independent variables included treatment, week, and the treatment-by-week interaction; subject served as a random effect; and the log transformed baseline daily hot flash severity score was used as a covariate; Test type: Superiority; p = 0.551, Repeated Measures Analysis of Covariance; Least Square Geometric Mean Ratio = 1.14, 95% CI 2-sided [0.74 to 1.74]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: A treatment-emergent adverse event is any adverse event that began or worsened after the initial dose of study drug and before the end of study.
  A serious adverse event is an adverse event that met at least 1 of the following serious criteria:
  * fatal
  * life threatening
  * required inpatient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect.
  * other medically important serious event A treatment-related adverse event (TRAE) is any treatment-emergent adverse event that per investigator review had a reasonable possibility of being caused by the study drug.
Time Frame: 16 weeks
Population: All participants who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 52 | 50
Participants
  Treatment-emergent adverse events (TEAEs) | 23 | 24
  Serious adverse events | 0 | 0
  TEAE leading to discontinuation of study drug | 0 | 0
  TEAE leading to discontinuation of study | 0 | 0
  Fatal adverse events | 0 | 0
  Treatment-related adverse events (TRAEs) | 5 | 3
  Treatment-related serious adverse events | 0 | 0
  TRAE leading to discontinuation of study drug | 0 | 0
  TRAE leading to discontinuation of study | 0 | 0
  Treatment-related fatal adverse events | 0 | 0

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of Erenumab After a Single Dose
Description: Blood samples were analyzed using an enzyme-linked immunosorbent assay (ELISA) following a validated analytical procedure.
Time Frame: Predose and 4 hours, 2, 3, 4, 8, 12, 15, 22, 29, 43, 50, 57, 64, 78, 85, and 113 days post-dose
Population: All participants who received erenumab and for whom at least 1 pharmacokinetic (PK) parameter or endpoint could be adequately estimated.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Erenumab
Number analyzed (Participants) | 50
μg/mL | 6.13 (2.86)

5. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Erunumab After a Single Dose
Time Frame: Predose and 4 hours, 2, 3, 4, 8, 12, 15, 22, 29, 43, 50, 57, 64, 78, 85, and 113 days post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Erenumab
Number analyzed (Participants) | 50
days | 7.0 [0.92 to 19]

6. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUClast) for Erenumab
Time Frame: Predose and 4 hours, 2, 3, 4, 8, 12, 15, 22, 29, 43, 50, 57, 64, 78, 85, and 113 days post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Erenumab
Number analyzed (Participants) | 50
day*μg/mL | 173 (84.6)

7. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) for Erenumab
Time Frame: Predose and 4 hours, 2, 3, 4, 8, 12, 15, 22, 29, 43, 50, 57, 64, 78, 85, and 113 days post-dose
Population: All participants who received erenumab and for whom at least 1 pharmacokinetic (PK) parameter or endpoint could be adequately estimated. AUCinf could not be accurately estimated for 23 participants who are excluded from the analysis.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Erenumab
Number analyzed (Participants) | 27
day*μg/mL | 190 (96.3)

8. Secondary Outcome: Terminal Half-life (T1/2) of Erenumab
Time Frame: Predose and 4 hours, 2, 3, 4, 8, 12, 15, 22, 29, 43, 50, 57, 64, 78, 85, and 113 days post-dose
Population: All participants who received erenumab and for whom at least 1 PK parameter or endpoint could be adequately estimated. T1/2 could not be accurately estimated for 23 participants who are excluded from the analysis. The terminal half-life calculated from this single dose study may not be representative of a clinically relevant half-life of erenumab.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Erenumab
Number analyzed (Participants) | 27
days | 12.1 (3.00)

9. Secondary Outcome: Number of Participants With Treatment-emergent Suicidal Ideation
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) was used to assess suicidal ideation during the study based on the following Yes/No questions:
  1. Have you wished you were dead or wished you could go to sleep and not wake up?
  2. Have you actually had any thoughts of killing yourself?
Time Frame: 16 weeks
Population: All participants who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 52 | 50
Participants | 0 | 0

10. Secondary Outcome: Number of Participants Who Developed Anti-erenumab Antibodies After a Single Dose
Description: Two validated assays were used to detect the presence of anti-erenumab antibodies. First, an electrochemiluminescent (ECL) bridging immunoassay was used to detect antibodies capable of binding erenumab. Second, a cell based bioassay was used to test positive binding antibody samples for neutralizing activity against erenumab.
  A participant was defined as positive for developing anti-erenumab antibodies if they were binding antibody positive postbaseline with a negative or no result at baseline. If a sample was positive for binding antibodies and demonstrated neutralizing activity at the same time point, the participant was defined as positive for neutralizing antibodies.
Time Frame: 16 weeks
Population: All participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 52 | 50
Participants
  Binding antibody positive | 0 | 5
  Neutralizing antibody positive | 0 | 4

ADVERSE EVENTS:
Time Frame: 16 Weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Erenumab 70 mg: Participants received a single dose of 70 mg erenumab administered by subcutaneous injection.
Arm/Group | Placebo | Erenumab 70 mg
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50
Other Adverse Events (participants affected / at risk) | 11/52 | 9/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | Erenumab 70 mg (N=50)
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.